CLINICAL TRIAL: NCT00754195
Title: Influence of Catheter Insertion Distance on the Quality of Thoracic Epidural Analgesia in the Context of Thoracotomy Procedures.
Brief Title: Insertion Distance of Thoracic Epidural Catheters in the Context of Thoracotomy Procedures.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08.071
Record Dates: First submitted 2008-09-15; First posted 2008-09-17 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Pain
Keywords: Thoracotomy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Insertion distance of thoracic epidural catheter: 3 cm
  Interventions: Other: Thoracic epidural catheter
- 2 (Active Comparator): Insertion distance of thoracic epidural catheter: 5 cm
  Interventions: Other: Thoracic epidural catheter
- 3 (Active Comparator): Insertion distance of thoracic epidural catheter: 7 cm
  Interventions: Other: Thoracic epidural catheter

INTERVENTIONS:
Other: Thoracic epidural catheter — Comparison of 3 insertion distances (3,5 and 7 cm) for a thoracic epidural catheter in the context of thoracic surgery.

SUMMARY:
This study is designed to compare thoracic epidural catheter insertion distances, in order to determine which is the best for pain relief following a thoracotomy.

HYPOTHESIS :

1. The quality of epidural analgesia upon coughing one hour following the end of surgery will not be inferior if the catheter is inserted 7 cm in the epidural space, versus 3 and 5 cm.
2. The quality of epidural analgesia upon coughing at 24 hour will not be inferior if the catheter is inserted 3 cm in the epidural space, versus 5 and 7 cm.

DETAILED DESCRIPTION:
Thoracic surgery such as posterolateral thoracotomy is associated with severe postoperative pain. Pain control is particularly important, as adequate analgesia allows rapid mobilisation and prevents complications related to immobility. Over the last years, thoracic epidural analgesia has become increasingly popular and is now considered the gold standard after thoracotomy. Thoracic epidural analgesia improves pain relief and also significantly decreases the incidence of morbidity and mortality following pulmonary resection. It also reduces the length of stay in the hospital and long-term pain 6 months after surgery. This method is now offered to a majority of patients undergoing a thoracotomy in our hospital.

The placement of a catheter in the thoracic epidural space remains a challenge for the anesthesiologist. Suboptimal placement of the catheter within the epidural space can result in inadequate pain relief. The distance at which the catheter must be advanced in the thoracic epidural space remains unknown. Insertion distance could influence the initial quality and distribution of sensory blockade, its duration, or both. Therefore, this study is designed to compare three catheter insertion distances, in order to help determine which is best for pain relief after a thoracotomy.

Methods :

1. Insertion of the epidural catheter :

   Patients will be randomly assigned to the following groups :
   * Group 1 : 3 cm insertion
   * Group 2 : 5 cm insertion
   * Group 3 : 7 cm insertion

   The anesthesiologist will insert the epidural catheter at T6-T7 before the induction of anesthesia for surgery. The usual medication will be used to make catheter installation comfortable. Standard non-invasive monitoring will be used.

   Correct placement of the epidural catheter will be assessed by infusing a bolus of 5 mL of lidocaine 1.5% with epinephrine 1 : 200,000. After induction of anesthesia and after placing the patient in the lateral decubitus position, the epidural infusion (bupivacaine 0.1% and fentanyl 2 mcg/mL) will be started at a rate of 0.1 mL/kg/h. Adjustments will be made between 4 to 16 mL/h with boluses of 0.1 mL/kg (maximum 7 mL) of solution as needed. Surgery will be performed under general anesthesia using a standardised protocol.
2. Post-operative analgesia :

   Pain will be assessed using a verbal numeric rating scale (NRS), where 0 refers to " no pain " and 10 refers to " the worst pain imaginable ". Pain at the surgical site and post-thoracotomy shoulder pain will be assessed separately. Post-thoracotomy shoulder pain will be treated with acetaminophen 975 mg every 6 hours and nonsteroidal antiinflammatory drugs (NSAIDs) or opioids as needed.

   Patients experiencing moderate to severe pain at the surgical incision site will receive a bolus of 0.1 mL/kg (maximum 7 mL) of epidural solution, and the infusion rate will be increased in 2 mL/h increments, to a maximum infusion rate of 16 mL/h. The infusion rate will be adjusted to maintain a pain score at the surgical site of 3 or less on the numeric rating scale. One hour after arrival in the recovery room, NRS during cough, at rest, and upon palpation, as well as loss of cold sensation will be assessed by a member of the research team who is blinded to the patient's group assignment. Total bupivacaine and morphine doses will be recorded.
3. Follow-up

At 24 hours after surgery, NRS during cough, at rest, and upon palpation, as well as loss of cold sensation, will be assessed by a member of the research team who is blinded to the patient's group assignment. Total bupivacaine and morphine doses will be recorded. Catheter distance at the skin will be verified for displacement.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older undergoing an elective thoracotomy.

Exclusion Criteria:

* Infection or sepsis
* Coagulopathy
* Hypovolemia
* Allergy to local anesthetics
* Neuropathy that could affect study assessments
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Quality of pain relief during cough | At one hour and 24 hours after surgery

SECONDARY OUTCOMES:
Quality of pain relief at rest | At one hour and 24 hours after surgery
Proportion of failed epidurals | At one hour and 24 hours after surgery
Wound palpation pain | At one hour and 24 hours after surgery
Loss of cold sensation around the wound | At one hour and 24 hours after surgery
Cumulative bupivacaine and morphine consumption | At one hour and 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Stephan R Williams, MD, PhD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (Hôpital Notre-Dame), Montreal, Quebec, Canada